CLINICAL TRIAL: NCT00080015
Title: A Phase II Open Label Study Investigating the Activity of Diflomotecan (BN80915) Administered at the Fixed Dose of 7mg as a 20 Minute Intravenous Infusion Once Every 3 Weeks in Patients With Sensitive Small Cell Lung Cancer (SCLC) Who Have Failed First-line Treatment With a Platinum Based Regimen.
Brief Title: Diflomotecan (BN80915) Administered Once Every 3 Weeks in Treating Patients With Sensitive Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-91-52990-708; 2004-001350-92 (EudraCT Number)
Record Dates: First submitted 2004-03-19; First posted 2004-03-23 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — diflomotecan

INTERVENTIONS:
Drug: Diflomotecan (BN80915)

SUMMARY:
This is a Phase II, open-label, multicenter, single-arm, exploratory "proof of concept" study. Diflomotecan (7 mg fixed dose) will be administered as a 20-minute IV infusion once every 3 weeks in patients with sensitive small cell lung cancer (SCLC) with progressive disease after first-line treatment with a platinum-based regimen.

ELIGIBILITY:
Main Inclusion Criteria:

* Documented small cell lung cancer (SCLC)
* Measurable disease
* One line of previous chemotherapy, including any platinum analogue, and excluding any camptothecin analogues, with objective response and relapsed no less than 3 months

Main Exclusion Criteria:

* Uncontrollable brain metastasis
* Treated with an investigational drug within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-03-12 (Actual); Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Overall objective response rate (tumour assessments should be performed every 6 weeks)

SECONDARY OUTCOMES:
Time to tumour progression
Time to treatment failure
Duration of overall response
Overall complete response, partial response and stable disease
Time to response
Six month and one year survival rates
Median survival
Best overall response
Overall objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen